CLINICAL TRIAL: NCT02193425
Title: Reliability Of The Human Brain Connectome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 140144; 14-AA-0144
Record Dates: First submitted 2014-07-16; First posted 2014-07-17 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Normal Physiology
Keywords: fMRI; Brain Connectivity; PET; 18FDG

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET FDG & MRI Scans (Experimental): The test-retest reproducibility of the gender and aging effects on FC measures (lFCD, C, L and S) acquired in RS and TS conditions.
  Interventions: Drug: F-18FDG; Device: MRI

INTERVENTIONS:
Drug: F-18FDG — 18F-Fluorodeoxyglucose (FDG)-PET session to assess the association between functional connectivity (FC) and glucose metabolism in the human brain.
Device: MRI — Two MRI/MRS sessions to evaluate test-retest reliability of functional connectivity (FC) at rest as well as during task performance.

SUMMARY:
Background:

- Magnetic resonance imaging (MRI) is used to investigate brain function. Researchers want to use MRI to better understand the function patterns and connections between brain regions in healthy people. This might help people with brain diseases in the future.

Objectives:

* To evaluate MRI methods performed twice on the same day.
* To evaluate brain function using positron emission tomography (PET).

Eligibility:

- Healthy volunteers at least 18 years old.

Design:

* Visit 1:
* Participants will be screened with medical history, physical exam, and interview about drug and alcohol use and psychiatric history.
* They will give blood and urine samples. Their breath will be tested for alcohol and smoking.
* Visit 2:
* Participants will have urine collected. They will have MRI scans, some while resting, some while doing tasks on a computer.
* The MRI scanner is a metal cylinder in a strong magnetic field. Participants will lie on a table that slides in and out of the cylinder, with a coil over their head. Participants will get earplugs for loud noises.
* Visit 3:
* Participants will have urine collected.
* A needle will guide a thin plastic tube (catheter) into each arm. The needle will be removed, leaving the catheter in the vein.
* Participants will then have a PET scan. They will get the chemical 18FDG in the catheter. They will lie on a bed that slides in and out of the PET scanner, with a cap on their head.
* Participants may have tests of memory, attention, concentration, and thinking. They may complete interviews, questionnaires, tests on paper or computer, and simple actions.
* Participants will wear a device for 1 week between visits to measure activity and sleep.

DETAILED DESCRIPTION:
Pr(SqrRoot)(Copyright)cis:

Objectives: The overarching goal of this study is to quantify the reproducibility of multiple measures of brain functional connectivity (FC) during resting conditions and during task performance. Secondary objectives are to assess the dynamic properties and energy requirements of the human brain connectome as well as the effects of physiologic noise, gender and aging on measures of brain functional connectivity at rest and during task performance.

Study population: 60 healthy males and 60 healthy females 18 years or older will be included.

Design: Participants will undergo two MRI/MRS sessions to evaluate test-retest reliability of FC at rest as well as during task performance, and one 18F-Fluorodeoxyglucose (FDG)-PET session to assess the association between FC and glucose metabolism in the human brain.

Outcome parameters: The variability of the gender and aging effects on FC measures (lFCD, L, C, and S) collected in RS and TS conditions , which will be quantified using volxelwise ICC (3,1). The variability of brain metabolite concentrations in precuneus.

ELIGIBILITY:
* INCLUSION CRITERIA:

All Participants:

* Older than 18 years of age.
* Ability to provide written informed consent as determined by physical examination and verbal communication. Capacity to consent will be determined by those obtaining the informed consent

EXCLUSION CRITERIA:

* Pregnant or breast feeding. Females of childbearing potential must have negative urine pregnancy test and not be currently breastfeeding. Post-menopausal or surgically sterile (tubal ligation or hysterectomy) females satisfy these criteria.
* The following current chronically used (within 2 months of study procedures) psychoactive medications or medications that can affect brain function (including but not limited to meperidine, tricyclic antidpressants, selective serotonin reuptake inhibitors (SSRIs), or serotonin norepinephrine reuptake inhibitors (SNRIs), stimulant or stimulant-like medications (amphetamine, methylphenidate, modafinil); opioid analgesics; antianginal agents; antiarrhythmics; systemic corticosteroids; anticholinergics; anticoagulants; anticonvulsants; antihistamines (sedating); beta blocker antihypertensives; antineoplastics; antiobesity; antipsychotics; anxiolytics

(benzodiazepine or barbiturates); lithium; muscle relaxants, and systemic steroids as determined by history and clinical exam.

* Current or past DSM-IV or DSM-5 diagnosis of a psychiatric disorder as determined by history and clinical exam including substance use disorder (except for nicotine/caffeine), alcoholism and alcohol dependence. Past history of a mental disorder as defined by DSM-IV or DSM-5 will be excluded only if it required hospitalization (any length), or chronic medication management (more than 4 weeks), and that could impact brain function at the time of the study.
* Those with a binge drinking history every month continuously for the last 10 years will also be excluded. Binge drinkers are those who being female consume 4 or more drinks and males consume 5 or more drinks in one occasion at least once a month.
* Major medical problems that can impact brain function at the time of the scan (including but not limited to HIV; central nervous system including seizures and psychosis; cardiovascular including hypertension and arrhythmias; metabolic, autoimmune, endocrine) as determined by history and clinical exam. Participants aged 60 and older with any medical problems that are controlled will not be excluded.
* Any clinically significant laboratory finding as determined during the screening procedures.
* Have had previous radiation exposure (from X-rays, PET scans, or other exposure) that, with the exposure from this study, would exceed NIH annual research limits.
* Head trauma with loss of consciousness for more than 30 minutes.
* Presence of ferromagnetic objects in the body that are contraindicated for MRI/MRS of the head (pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments), fear of enclosed spaces, or other standard contraindication to MRI/MRS (self-report checklist).
* Cannot lie comfortably flat on back for up to 2 hours in the PET and MRI/MRS scanners.
* Body weight > 250 kg. This is the upper limit that the bed of the MR scanner can accommodate.
* NIH employees who are study investigators, as well as their superiors, subordinates and immediate family members (adult children, spouses, parents, siblings).
* Non-English speakers (subjects must be able to read and comprehend English).

  * Subjects will not be excluded from enrollment onto this study if their urine test is positive for drugs. However, if they test positive on scheduled study procedure days involving study imaging (MRI/MRS and PET) and Neuropsychological testing, the procedures will be postponed and rescheduled. We will allow for up to 3 rescheduled study days that were the result of positive urine drug screens. If the drug test is positive on the third rescheduled visit, the participant will be withdrawn from the study.

The intent of the research has no prospect of direct benefit to the subject. Therefore, we are excluding non-English speakers in this research study since it includes the administration of questionnaires, surveys and assessments that are validated for English, although some are available in Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-06-08 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
The overarching goal of this study is to quantify the reproducibility of multiple measures of brain functional connectivity (FC) during resting conditions and during task performance. | end of study
  The test-retest reproducibility of the gender and aging effects on FC measures (lFCD, C, L and S) acquired in RS and TS conditions.

SECONDARY OUTCOMES:
The correlation between glucose metabolism, CBF, lFCD, C, L and S and its contribution to between- subjects FC-variability during RS. | end of study
  To assess the dynamic properties and energy requirements of the human brain connectome as well as the effects of physiologic noise, gender and aging on measures of brain functional connectivity at rest and during task performance.
The association between IFCD and the underlying structural connectivity and its contribution to between- subjects FC-variability during RS. | end of study
  To assess the dynamic properties and energy requirements of the human brain connectome as well as the effects of physiologic noise, gender and aging on measures of brain functional connectivity at rest and during task performance
The correlation between physiologic noise and FC measures (lFCD, C, L and S) and its contribution to within- subjects FC-variability during RS and TS conditions. | end of study
  To assess the dynamic properties and energy requirements of the human brain connectome as well as the effects of physiologic noise, gender and aging on measures of brain functional connectivity at rest and during task performance
The dynamics of the FC measures (lFCD, C, L and S) and its contribution to within- subjects FC-variability during RS and TS conditions. | end of study
  To assess the dynamic properties and energy requirements of the human brain connectome as well as the effects of physiologic noise, gender and aging on measures of brain functional connectivity at rest and during task performance

CONTACTS AND LOCATIONS:
Overall Officials: Dardo G Tomasi, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Data is analyzed in groups so no individual information will be shared.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-AA-0144.html